CLINICAL TRIAL: NCT00509340
Title: Cognitive Behavioral Adherence Intervention for Depressed HIV Patients
Brief Title: Cognitive Behavioral Therapy to Help HIV Infected Adults With Depression to Adhere to Antiretroviral Therapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Inability to recruit enough eligible participants at study site.
Sponsor: RAND (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Glenn Wagner, Senior Behavioral Scientist, RAND
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R34MH077503 (NIH); R34MH077503 (NIH); DAHBR 9A-ASNM
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Depression; HIV Infection
Keywords: antiretroviral; adherence; poor antiretroviral adherence
MeSH Terms: conditions — Depression; HIV Infections | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Participants will receive usual clinical care, which may or may not include mental health treatment
- 2 (Experimental): Participants will receive cognitive behavioral intervention
  Interventions: Behavioral: Cognitive behavioral therapy (CBT)

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy (CBT) — Participants in this group will receive individual sessions of cognitive-behavioral training for improvement of medication adherence and reduction of depression.
  Arms: 2

SUMMARY:
This study will compare the effectiveness of a cognitive behavioral intervention versus usual clinic care in helping HIV infected adults with depression to take their HIV medications on schedule.

DETAILED DESCRIPTION:
Antiretroviral therapy (ART) is a type of medication treatment for HIV that impairs the virus's ability to multiply. When used properly, it has been shown to be successful in reducing HIV-related deaths. A high adherence rate to ART is required to adequately suppress the virus, limit drug resistance, and reduce transmission. HIV infected people who are depressed often experience increased difficulty with adhering to their ART regimen. This study will compare the effectiveness of a cognitive behavioral intervention that targets both depression and adherence versus usual care practices which may or may not include mental health intervention with the goal of improving ART adherence among HIV infected adults with depression who are experiencing difficulty with adhering to their medication regimen.

This study will last 24 weeks. Participants will be randomly assigned to receive the cognitive behavioral intervention or usual care. Study visits for all participants will occur at baseline and Weeks 4, 8, 16, and 24. Those receiving the intervention will also have visits at Weeks 1 and 2. Participants receiving the intervention will attend five individual treatment sessions followed by one to three booster treatment sessions; these sessions will coincide with the study visits.

ELIGIBILITY:
Inclusion Criteria:

* reports significant depressive symptoms as indicated by score of 10 or greater on PHQ-9
* Currently taking ART for HIV infection
* Less than 90% adherence rate to ART regimen
* Capable of walking and in stable health
* Speaks fluent English

Exclusion Criteria:

* Depression therapy is needed immediately
* Meets criteria for current drug dependency
* Current diagnosis of psychotic disorder or bipolar depression

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2007-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Microelectronic medication adherence | Measured at Weeks 16 and 24

SECONDARY OUTCOMES:
Self-reported depression | Measured at Weeks 16 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Glenn J. Wagner, PhD, Principal Investigator — RAND
Locations (1):
- LA Biomedical Institute at Harbor-UCLA, Torrance, California, United States